CLINICAL TRIAL: NCT01018446
Title: Determination of Optimal Busulfan Dose Using Pharmacokinetic Modeling in Hematopoietic Stem Cell Transplantation
Brief Title: Hematopoietic Stem Cell Transplantation Based on Pharmacokinetic and Pharmacodynamic Modeling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Korea National Enterprise for Clinical Trials, Korea National Enterprise for Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-SCT-0802
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic stem cell transplantation with busulfan based conditioning
MeSH Terms: interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan, Pharmacokinetic (Experimental): To develop a method to determine optimal dose of busulfan through pharmacokinetic study in hematopoietic stem cell transplantation.
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — First dose: busulfan (120 mg/m2 ivs once daily) (if age<1 yr: 80 mg/ m2) Second to forth dose: according to the daily pharmacokinetic study

SUMMARY:
In this study the investigators plan to develop a method to determine optimal busulfan dose through pharmacokinetic study.

DETAILED DESCRIPTION:
Busulfan is a highly toxic drug with narrow therapeutic window used for the conditioning of hematopoietic stem cell transplantation. High exposure is associated with systemic toxicity such as veno-occlusive disease (VOD) and underexposure is associated with graft failure or relapse. In this study we plan to develop a method to determine optimal busulfan dose through pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

1. Hematopoietic stem cell transplantation with busulfan based conditioning
2. Age: no limits.
3. Performance status: ECOG 0-2.
4. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases. 1. Heart: a shortening fraction > 30% and ejection fraction > 45%. 2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal. 3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
5. Patients must lack any active viral infections or active fungal infection.
6. Appropriate donor is available: Matched in 6/6 of A, B, DR loci.
7. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To develop a method to determine optimal dose of busulfan through pharmacokinetic study in hematopoietic stem cell transplantation. | For 4 days used Buslufan through pharmacokinetic study in hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
To evaluate survival, toxicities, engraftment rate of patients received optimal dose of busulfan. | 1, 3, 6 and 12 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehangno, Jongno-gu, South Korea